CLINICAL TRIAL: NCT07260357
Title: Comparison Of Clinical And Radiological Success Of Pulpotomy Treatments Performed With Proroot MTA, NeoPUTTY MTA, TheraCal PT In Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: necmettin erbakan university Scientific Research Projects (BAP) (Unknown)
Responsible Party: Principal Investigator, Halenur Altan, Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NecmettinEU03
Record Dates: First submitted 2025-07-15; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Dentin Caries
Keywords: Pulpotomy; Primary Teeth; Mineral Trioxide Aggregate

STUDY DESIGN:
Intervention Model Description: Treatment selection of patients meeting the inclusion criteria was made using the randomized sealed envelope method. One envelope was created for each group and the patient was asked to choose which pulpotomy material would be used before the procedure. The procedure was performed by a single researcher (M.T.) who was receiving specialist training in pediatric dentistry. The teeth were restored with stainless steel crowns after the amputation treatment. Intraoral photographs were taken from the patients at the beginning, after cavity preparation and after the restoration was completed, and periapical radiographs were taken after the restorations were completed to control the restorations. The patients were called for control sessions at 6 and 9 months. A maximum of one periapical radiograph was taken from each tooth. The teeth were checked by 2 physicians (M.T. and H.A.) and recorded in the case report forms according to the determined clinical and radiographic evaluation criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ProRoot MTA White (Tulsa Dental Products, Tulsa, USA) (Experimental): Pro Root MTA Root Canal Repair Material
  Interventions: Other: ProRoot MTA Pulpotomy
- NeoPUTTY (NuSmile, Houston, USA) (Experimental): Next Generatıon Pre-Mıxed Root & Pulp Treatment Materıal
  Interventions: Other: NeoPUTTY MTA Pulpotomy
- ThraCal PT (Bisco Dental Products, Schaumburg IL, Amerika) (Experimental): BISCO's TheraCal PT is a dual-cured, resin-modified calcium silicate pulpotomy treatment.
  Interventions: Other: TheraCal PT Pulpotomy

INTERVENTIONS:
Other: ProRoot MTA Pulpotomy — Teeth were pulpotomized with Pro-Root MTA in this group.
  Arms: ProRoot MTA White (Tulsa Dental Products, Tulsa, USA)
Other: NeoPUTTY MTA Pulpotomy — Teeth were pulpotomized with Neo-Putty MTA in this group.
  Arms: NeoPUTTY (NuSmile, Houston, USA)
Other: TheraCal PT Pulpotomy — Teeth were pulpotomized with Theracal PT in this group.
  Arms: ThraCal PT (Bisco Dental Products, Schaumburg IL, Amerika)

SUMMARY:
The goal of this randomized clinical trial is to compare clinical and radiological success rates of NeoPutty MTA, ProRoot MTA and TheraCal PT pulpotomy in 4-10 years old healthy pediatric patients. The main question it aims to answer is:

Which of these 3 materials are best suited for pulpotomy treatment in the aspect of clinical and radiological success rates.

Participants will undergo a pulpotomy treatment in primary molar teeth with one of these materials used.

DETAILED DESCRIPTION:
This study was conducted on primary molar patients who applied to Necmettin Erbakan University Faculty of Dentistry Department of Pedodontics for a routine check-up, did not have any systemic problems, had a score of 3 and 4 according to the Frankl Behavior Scale, and whose parents' approval could be obtained, and had a pulp-related and active caries appearance in the lower jaw. Patients between the ages of 4 and 10 who are indicated for dental pulpotomy treatment will be included.

In our prospective randomized clinical study;

Pulpotomy treatment; Infiltrative/mandibular anesthesia is applied to the primary lower molar teeth, which are in contact with the pulp and have not experienced spontaneous pain, and wait until numbness occurs. Under rubber dam isolation, soft caries in the lower primary molar tooth is removed with a steel round bur.

Removal of pulp tissue: Starting from where the pulp is exposed, 1-2 mm is removed with a water-cooled high-speed diamond round bur.

Bleeding Control: It is washed with sterile serum and the cavity is disinfected using a cotton pellet impregnated with 2.5% Sodium Hypochlorite. It is checked that there is no residual pulp tissue left. For hemostasis, a cotton pellet impregnated with physiological saline is placed in the cavity.

Control group (Pro Root MTA) Pro Root MTA consists of powder and liquid components. The liquid part is added to the powder, mixed and placed in 30 primary molars as pulpotomy material. Glass ionomer cement is placed on it as a base material and the treatment is completed by making a permanent restoration with a stainless steel crown.

Working group (NeoPUTTY MTA) NeoPUTTY MTA is in injector form and has a paste consistency. Taken using a hand tool It is placed in 30 primary molars as pulpotomy material. As a base material on it Glass ionomer cement is placed and the treatment is completed by making a permanent restoration with a stainless steel crown.

Study group (Theracal PT) Theracal PT is in the form of a resin-containing syringe and is applied directly to 30 primary molars as pulpotomy material and polymerized with the help of a radiation device. Glass ionomer cement is placed on it as a base material and the treatment is completed by making a permanent restoration with a stainless steel crown.

When the literature is examined within the scope of our research, there are a limited number of studies comparing Pro Root MTA with NeoPUTTY MTA and Theracal PT. In this thesis study, it was aimed to compare its success on the pulp with the materials in the study group by using Pro Root MTA, which has proven its success on the pulp in the literature, in the control group. After the treatment of the teeth is completed, participants will be called for 6th and 9th month checks. During the control sessions, clinical and radiological evaluations of the relevant teeth will be made and periapical radiographs will be taken, maximum one from each tooth.

ELIGIBILITY:
Inclusion Criteria:

* Primary molars with active caries and pulp exposure, assessed after intraoral periapical radiograph examination
* Presence of pulp exposure during caries excavation
* More than two-thirds of root length present
* No history of spontaneous pain
* Children aged 4-10 years with Frankl's positive or definitely positive behavior

Exclusion Criteria:

* Teeth with internal or external root resorption, periapical lesions, or widening of the periodontal ligament (PDL)
* Presence of sinus tracts or history of swelling
* Uncontrolled pulpal bleeding from the tooth, even after 5 minutes
* No pulp exposure during caries excavation
* Patients or parents unwilling to participate in the study

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical Success Of Pulpotomy Treatments Performed With Proroot MTA, NeoPUTTY MTA, TheraCal PT In Primary Teeth | 6 months and 9 months post-treatment
  Clinical success will be evaluated at 6- and 9-month follow-up examinations by assessing the following parameters: spontaneous pain, tenderness to percussion, swelling, sinus/fistula formation, and pathological mobility.
  Each parameter will be recorded as positive (present) or negative (absent). Tooth mobility will be graded according to Miller's Mobility Classification (Grades 0-3).
  A tooth will be considered clinically successful if all parameters are negative (no symptoms) and mobility is within Miller's Grade 0-1.
  Data will be aggregated and reported as the number and percentage of teeth with clinical success for each pulpotomy material group (ProRoot MTA, NeoPUTTY, and TheraCal PT).
Clinical And Radiological Success Of Pulpotomy Treatments Performed With Proroot MTA, NeoPUTTY MTA, TheraCal PT In Primary Teeths | 6 months and 9 months post-treatment
  Radiographic success will be evaluated at 6- and 9-month follow-up visits using standardized periapical radiographs. Each radiograph will be examined for the presence or absence of the following findings: periapical radiolucency, furcal involvement, internal or external root resorption, and widening of the periodontal ligament space.
  Each parameter will be recorded as positive (absent pathology) or negative (presence of any pathology).
  Teeth showing no pathological findings (i.e., all parameters positive) will be classified as radiographically successful, whereas those showing any pathological change (negative) will be classified as radiographic failures.
  Evaluations will be performed independently by two blinded examiners. Data will be aggregated and reported as the number and percentage of radiographically successful teeth for each pulpotomy material group (ProRoot MTA, NeoPUTTY, and TheraCal PT).

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Faculty of Dentistry, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will share the results.

REFERENCES:
- [Background] Bossu M, Iaculli F, Di Giorgio G, Salucci A, Polimeni A, Di Carlo S. Different Pulp Dressing Materials for the Pulpotomy of Primary Teeth: A Systematic Review of the Literature. J Clin Med. 2020 Mar 19;9(3):838. doi: 10.3390/jcm9030838. PMID 32204501